CLINICAL TRIAL: NCT06995469
Title: Efficacy of a Passive Lower Limb Exoskeleton on Plantar Pressure Distribution to Reduce on Plantar Pressure Distribution to Reduce Prolonged Standing Injuries: Prolonged Standing Injuries
Brief Title: Efficacy of a Passive Lower Limb Exoskeleton in Reducing Plantar Pressure and Injuries From Prolonged Standing
Acronym: PELLEPSI
Status: Completed | Type: Observational
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Principal Investigator, Javier Ferrer Torregrosa, HEAD OF PODIATRY DEPARTMENT, Fundación Universidad Católica de Valencia San Vicente Mártir
Other Study IDs: UCV/2024-2025/030
Record Dates: First submitted 2025-05-06; First posted 2025-05-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Health-Related Behavior
Keywords: Passive exoskeleton; Lower limbs; Prolonged standing; Plantar pressure; Occupational ergonomics
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exoskeleton: This single-group cohort consists of participants assessed under two conditions: (1) performing prolonged standing tasks with the use of a passive lower-limb exoskeleton (Chairless Chair® 2.0) and (2) performing the same tasks without the exoskeleton.
  Each participant serves as their own control in a within-subject, repeated-measures design to evaluate changes in plantar pressure distribution, postural stability, perceived fatigue, and device usability.
  Interventions: Procedure: Chairless Chair® 2.0 Passive Lower-Limb Exoskeleton

INTERVENTIONS:
Procedure: Chairless Chair® 2.0 Passive Lower-Limb Exoskeleton — Participants used a passive lower-limb exoskeleton (Chairless Chair® 2.0) during their regular work tasks involving prolonged standing. The device enables a semi-seated posture without the need for external power, aiming to reduce lower limb strain.
  The intervention involved each participant performing their typical standing tasks once with the exoskeleton and once without it, in a within-subject repeated-measures design. Each participant served as their own control.
  Objective data were collected using a plantar pressure platform (Podoprint S4, Namrol) to measure:
  Plantar pressure distribution
  Postural stability
  Body sway

SUMMARY:
This quasi-experimental study evaluates the effectiveness of a passive lower-limb exoskeleton (Chairless Chair® 2.0) in redistributing plantar pressure and reducing injuries caused by prolonged standing in workplace settings. Conducted on 25 participants, the research measured plantar pressure, body sway, and postural stability with and without the exoskeleton using a pressure platform. Additionally, user fatigue and satisfaction were assessed through validated questionnaires (Borg CR10, QUEST 2.0). The results aim to determine the device's preventive potential regarding musculoskeletal and circulatory issues, contributing to improved ergonomic health and work performance.

DETAILED DESCRIPTION:
Prolonged standing is a common requirement in various professional sectors (e.g., healthcare, industry), and is associated with increased risks of musculoskeletal and circulatory disorders, especially in the lower limbs. Conditions such as plantar fasciitis, chronic venous insufficiency, and pressure ulcers are prevalent. These affect worker health, comfort, and productivity, and impose economic burdens on employers and healthcare systems.

Objective To evaluate the effectiveness of a passive exoskeleton for the lower limbs (Chairless Chair® 2.0) in redistributing plantar pressure and reducing musculoskeletal injuries associated with prolonged standing. The study also investigates the device's influence on postural stability, perceived fatigue, and user comfort.

Methodology Study design: Quasi-experimental with repeated measures (participants act as their own control).

Participants: 25 adult workers (aged 18-60), with ≥6 months of exposure to prolonged standing at work. Exclusion criteria included pre-existing musculoskeletal or circulatory disorders and use of orthopedic devices.

Device: Chairless Chair® 2.0 by Noonee Germany GmbH-a passive, non-powered exoskeleton enabling users to alternate between standing and semi-sitting positions.

Tools and Measurements:

Podoprint S4 pressure platform to measure:

Plantar pressure distribution (forefoot, midfoot, heel)

Body sway and stability (center of pressure displacement)

CR10 Borg scale for fatigue

QUEST 2.0 for usability and satisfaction

Data Analysis:

Quantitative analysis using SPSS and JASP

Paired t-tests or Wilcoxon tests for comparisons

Spearman correlations and Chi-square tests for categorical relationships

Statistical significance set at p < 0.05

Key Variables Dependent: Plantar pressure (kPa), body sway (cm²), postural stability (mm/s), fatigue perception, comfort.

Independent: Use of exoskeleton, age, gender, BMI, type of footwear, reported discomfort.

Ethical and Legal Framework Ethical approval granted by the Comité de Ética de la Universidad Católica de Valencia (CEI).

Compliance with LOPDGDD, GDPR, and Declaration of Helsinki.

Informed consent obtained; anonymity and data protection were strictly maintained.

Expected Outcomes Reduction in peak plantar pressure and postural sway when using the exoskeleton.

Improvement in stability and fatigue levels.

Enhanced user comfort and satisfaction, making the device a feasible ergonomic intervention.

Significance This study seeks to fill a gap in scientific literature regarding the biomechanical benefits of passive lower-limb exoskeletons in real work environments, providing evidence for their role in injury prevention, ergonomic improvement, and worker well-being.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 60 years

Currently employed in jobs requiring prolonged standing (≥4 hours/day)

Minimum 6 months of work experience in such standing-intensive roles

Physically capable of performing normal job tasks

Able and willing to provide informed consent

Exclusion Criteria:

Diagnosis of musculoskeletal or circulatory conditions (e.g., plantar fasciitis, varicose veins, chronic venous insufficiency)

Current use of orthopedic or ergonomic devices, such as foot orthoses

Uncontrolled medical conditions that may pose a risk (e.g., uncontrolled hypertension)

Pregnancy

Inability to understand or comply with study procedures

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study population consists of adults aged 18-65 who work in roles requiring ≥4 hours of standing daily, with at least 6 months of continuous experience. Participants were selected through purposive sampling based on specific inclusion/exclusion criteria. Individuals with diagnosed musculoskeletal or circulatory disorders or those already using orthopedic/ergonomic devices were excluded. This group reflects a real-world ergonomic risk population, suitable for assessing the preventive efficacy of a passive lower limb exoskeleton in the workplace.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Plantar Pressure Distribution With vs. Without Passive Exoskeleton Use Change in Plantar Pressure Distribution With vs. Without Passive Exoskeleton Use Change in Plantar Pressure Distribution With vs. Without Passive Exoskeleton Use | Immediately after task performance in each condition (with and without exoskeleton) - approximately same workday or within 1-2 days
  Mean plantar pressure values (in kilopascals, kPa) will be measured in key foot regions (heel, midfoot, forefoot) using the Podoprint S4 platform. Data will be collected under two conditions: while performing tasks with the Chairless Chair® 2.0 and without it. The comparison will assess the exoskeleton's effectiveness in redistributing plantar loads during prolonged standing.

SECONDARY OUTCOMES:
Change in Postural Stability With vs. Without Passive Exoskeleton | Immediately after task performance in each condition (with and without exoskeleton)
  Postural stability and center of pressure (COP) displacement (in cm² and mm/s) will be measured during static standing using the Podoprint S4 pressure platform. The goal is to evaluate whether the exoskeleton improves balance and reduces body sway during prolonged standing tasks.
Perceived Fatigue After Work Tasks With vs. Without Exoskeleton | Immediately after task completion in each condition - within same workday
  Fatigue in the lower extremities will be assessed using the Borg Scale CR10, a validated ordinal questionnaire ranging from 0 (no exertion) to 10 (maximum exertion). A higher score indicates greater perceived fatigue. Participants will report their perception of exertion immediately after completing the tasks, both with and without the exoskeleton.
User Comfort and Usability of the Passive Exoskeleton | After using the exoskeleton during a full work session - within 1 day
  Participants will complete the QUEST 2.0 (Quebec User Satisfaction Evaluation of Assistive Technology) questionnaire, which includes scores on a scale from 1 (very dissatisfied) to 5 (very satisfied). Higher scores reflect greater satisfaction and positive perception of the comfort, usability and acceptability of the device. The results will allow assessment of the practical acceptability of the exoskeleton in real work environments.

CONTACTS AND LOCATIONS:
Overall Officials: JAVIER FERRER TORREGROSA, Dr., Principal Investigator — UNIVERSIDAD CATOLICA DE VALENCIA
Locations (1):
- Clinicas UCV, Valencia, València, Spain

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be made publicly available through publication in a peer-reviewed scientific journal and presentation at academic conferences. A summary of the findings will also be provided to participants upon request. In addition, anonymized datasets and key outcome summaries may be shared for academic and research purposes.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: All published results and associated materials will be accessible indefinitely through institutional repositories or journal archives
Access Criteria: Open access

REFERENCES:
- [Background] Liu L, Wei W, Zheng K, Diao Y, Wang Z, Li G, Zhao G. Design of an Unpowered Ankle-Foot Exoskeleton Used for Walking Assistance. Annu Int Conf IEEE Eng Med Biol Soc. 2021 Nov;2021:4501-4504. doi: 10.1109/EMBC46164.2021.9630707. PMID 34892218
- [Background] Steinhilber B, Seibt R, Rieger MA, Luger T. Postural Control When Using an Industrial Lower Limb Exoskeleton: Impact of Reaching for a Working Tool and External Perturbation. Hum Factors. 2022 Jun;64(4):635-648. doi: 10.1177/0018720820957466. Epub 2020 Sep 28. PMID 32988243
- [Background] Kong YK, Park CW, Cho MU, Kim SY, Kim MJ, Hyun DJ, Bae K, Choi JK, Ko SM, Choi KH. Guidelines for Working Heights of the Lower-Limb Exoskeleton (CEX) Based on Ergonomic Evaluations. Int J Environ Res Public Health. 2021 May 13;18(10):5199. doi: 10.3390/ijerph18105199. PMID 34068352